CLINICAL TRIAL: NCT00864136
Title: MiCo - Mirena or Conventional Medical Treatment for Menorrhagia
Brief Title: Mirena or Conventional Medical Treatment for Menorrhagia
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 14697; MA0701 (Other: Company Internal); MA0901 - non-East Asia (Other: Company Internal)
Record Dates: First submitted 2009-03-17; First posted 2009-03-18 (Estimated); Last update posted 2015-07-01 (Estimated); Status verified 2015-06

CONDITIONS: Menorrhagia
MeSH Terms: conditions — Menorrhagia | interventions — Levonorgestrel

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Group 1
  Interventions: Drug: Levonorgestrel (Mirena, BAY86-5028)
- Group 2
  Interventions: Drug: Conventional medical treatment
- Group 3
  Interventions: Drug: Conventional medical treatment

INTERVENTIONS:
Drug: Levonorgestrel (Mirena, BAY86-5028) — Women using Mirena for treatment of menorrhagia
  Groups: Group 1
Drug: Conventional medical treatment — Women using combined oral contraceptives, oral/injectable progestogens, non-steroidal anti-inflammatory drug
  Groups: Group 2
Drug: Conventional medical treatment — Women using anti-fibrinolytic agent for treatment of menorrhagia
  Groups: Group 3

SUMMARY:
The aim of this prospective, non-interventional post-marketing surveillance study is to obtain data on safety and efficacy of Mirena in treatment of prolonged or heavy menstrual bleeding (Menorrhagia) under daily-life treatment conditions.

It is planned to conduct the study in about 10 countries with a total of 1000 patients. In several countries, a comparator group will also be documented.

For each patient, an initial visit and one to three follow-up visits after about 3, 6 and 12 months will be documented by the treating physician on the case report form. Observations include the patient's demographic parameters (date of birth, height, weight, race and smoking habits), previous contraceptives and menorrhagia treatment, gynaecological history, baseline menstruation, result of insertion, concomitant medications and diseases as well as menorrhagia symptoms. Overall treatment success will be evaluated at the end of treatment including number of weeks until improvement and reduction of menstrual bleeding with respect to duration and severity, and patient's satisfaction.

DETAILED DESCRIPTION:
The "MiCo - Mirena or conventional medical treatment for menorrhagia" study consist of two parts, MiCo Asia-Pacific and MiCo MA0901 (Rest of World).

Data from both parts will be analysed in separate pools as well as in a global pool. The trial alias are IMPACT Nos. 14697, 14536 (NCT01085487).

ELIGIBILITY:
Inclusion Criteria:

* Women between the ages of 18-45 (inclusive) not intending to get pregnant during the next year
* Women complaining of heavy menstrual bleeding over several consecutive cycles
* Women without structural or histological abnormality of the uterus, or with fibroids less than 3 cm in diameter which are causing no distortion of the uterine cavity (eligible for pharmaceutical treatment according to the NICE guideline 2007)
* Informed consent (where required by laws or regulations)

Exclusion Criteria:

* The contraindications and warnings of the respective Summary of Product Characteristics (Mirena, combined oral contraceptives, oral/injectable progestogens, non-steroidal anti-inflammatory drug, or anti-fibrinolytic agent) must be followed.
* Women taking hormone replacement therapy
* Women with symptoms such as intermenstrual or post-coital bleeding, unless an endometrial biopsy has been performed and pathology excluded
* Women with fibroids that are palpable abdominally or who have intra-cavity fibroids and/or whose uterine length as measured at ultrasound or hysteroscopy is greater than 12 cm (NICE guideline 2007)
* Women on anticoagulative therapy or other treatment (including e.g. Copper IUD use) known to cause menorrhagia

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women with a diagnosis of idiopathic menorrhagia can be enrolled after decision for treatment has been made.
Sampling Method: Non-Probability Sample
Enrollment: 647 (Actual)
Dates: Start 2008-11; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Cumulative continuation rate stratified by history of previous treatment(s) for menorrhagia | at 12 months

SECONDARY OUTCOMES:
Bleeding pattern | at 12 months
Patient satisfaction at end of documentation | at 12 months
Impact of the therapy in terms of patient-derived health outcomes (validated patient questionnaire) | at 12 months
Adverse events collection | at 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (8):
- Many Locations, China
- Many Locations, Hong Kong
- Many Locations, Indonesia
- Many Locations, Malaysia
- Many Locations, Pakistan
- Many Locations, South Korea
- Many Locations, Taiwan
- Many Locations, Thailand

REFERENCES:
- [Derived] Lee BS, Ling X, Asif S, Kraemer P, Hanisch JU, Inki P. Levonorgestrel-releasing intrauterine system versus conventional medical therapy for heavy menstrual bleeding in the Asia-Pacific region. Int J Gynaecol Obstet. 2013 Apr;121(1):24-30. doi: 10.1016/j.ijgo.2012.10.028. Epub 2013 Jan 20. PMID 23340271